CLINICAL TRIAL: NCT03780868
Title: External Dacryocystorhinostomy Versus Canalicular Silicone Intubation With Mitomycin C in Primary Acquired Nasolacrimal Duct Obstruction
Brief Title: External DCR Versus Canalicular SI With MMC in NLDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Amin Faisal Ellakwa, assistant professor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ebsar ophthalmic Center
Record Dates: First submitted 2018-12-09; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Primary Acquired Nasolacrimal Duct Obstruction
Keywords: External DCR, canalicular silicone intubation, Mitomycin C

STUDY DESIGN:
Intervention Model Description: compare external dacryocystorhinostomy versus canalicular silicone intubation with the use of Mitomycin C (MMC) in primary acquired nasolacrimal duct obstruction (NLDO).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- external DCR (Active Comparator): A curvilinear incision of 10-15 mm length was made along the anterior lacrimal crest .
  The smaller end of the blunt dissector was used to fracture Lamina papyracea, the parchment like bone of the posterior half of the lacrimal fossa. the nasal mucosa was stripped from lacrimal bone with the help of Traquair's periosteal elevator, An osteotomy of approximately 12.5 x10mm was created with successive punching of bone by Cittelli's punch. Lacrimal sac and nasal mucosa were opened in a 'H' fashion with the no.11 Bard-Parker blade and Bowman's probe was in place, to form a large anterior and smaller posterior flap.
  Interventions: Procedure: external dacryocystorhinostomy; Procedure: canalicular silicone intubation with MMC
- silicone intubation with MMC (Active Comparator): Bowman's probe was gently inserted into the inferior canalicular system, until a hard stop was felt in the lacrimal sac, after which it was rotated into the NLD to reach below the inferior concha. The probe was then withdrawn via the inferior punctum and the process was repeated for the upper canaliculus.
  After irrigation with normal saline to confirm duct patency, irrigation was performed by introducing 1 ml of MMC (0.5 mg/ml) into the duct with a syringe, the ocular surface then irrigatedby normal saline. Intubation was done by a silicone tube connected by each of its end to a malleable steel guide. A grooved director was placed under the inferior turbinate to guide the probe out of the nose, after which the steel guide was cut from the silicone tube
  Interventions: Procedure: external dacryocystorhinostomy; Procedure: canalicular silicone intubation with MMC

INTERVENTIONS:
Procedure: external dacryocystorhinostomy — external DCR under general anesthesia with standard sterilization procedures.
Procedure: canalicular silicone intubation with MMC — canalicular silicone intubation with MMC under general anesthesia with standard sterilization procedures.

SUMMARY:
While external DCR is the gold standard procedure for primary NLDO as well as complicated cases, SI with MMC could achieve comparable success rates in primary acquired NLDO, hence should be considered as an alternative as a safe and minimally invasive procedure.

DETAILED DESCRIPTION:
Purpose: To compare external dacryocystorhinostomy versus canalicular silicone intubation with the use of Mitomycin C (MMC) in primary acquired nasolacrimal duct obstruction (NLDO).

Methods: the study was carried out at the department of Ophthalmology, Menoufia university Hospital, Egypt, between June 2012 to July 2014. Fifty-six patients who were diagnosed with primary acquired NLDO. Patients were randomly allocated into two groups: thirty cases underwent external DCR and twenty-six cases underwent silicone intubation with MMC.

ELIGIBILITY:
Inclusion Criteria:

* primary acquired NLDO

Exclusion Criteria:

* All other secondary causes of NLDO

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2014-07-31 (Actual)

PRIMARY OUTCOMES:
external DCR | 2 years
  patency of lacrimal passage was tested by height of tear meniscus and lacrimal syringing. On the basis of subjective and objective evaluation, patients were categorized into three groups: successful surgery (asymptomatic, normal tear meniscus and patent lacrimal system with syringing procedure), improvement (watery eye and/or discharge, moderate tear meniscus and partially patent lacrimal system with syringing procedure with mild regurgitation from the puncta) and failed surgery (watery eye and/or discharge, high tear meniscus and non-patent lacrimal system).

OTHER OUTCOMES:
canalicular silicone intubation with MMC | 2 years
  patency of lacrimal passage was tested by height of tear meniscus and lacrimal syringing. On the basis of subjective and objective evaluation, patients were categorized into three groups: successful surgery (asymptomatic, normal tear meniscus and patent lacrimal system with syringing procedure), improvement (watery eye and/or discharge, moderate tear meniscus and partially patent lacrimal system with syringing procedure with mild regurgitation from the puncta) and failed surgery (watery eye and/or discharge, high tear meniscus and non-patent lacrimal system).

IPD SHARING:
Plan to Share IPD: No